CLINICAL TRIAL: NCT03902795
Title: Functional and Morphological Results of macula-on and Macula-off Rhegmatogenous Retinal Detachment Treated With Pars Plana Vitrectomy and Sulfur Hexafluoride Gas Tamponade
Brief Title: Functional and Morphological Results of Rhegmatogenous Retinal Detachment Treated With Vitrectomy
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: 0004
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Retinal Detachment; Vitrectomy
Keywords: Rhegmatogenous retinal detachment; Vitrectomy; Metamorphopsia; M-charts; Microperimetry
MeSH Terms: conditions — Retinal Detachment; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of 62 eyes: Group of 62 eyes with rhegmatogenous retinal detachment who underwent successful vitrectomy with SF6 tamponade
  Interventions: Diagnostic Test: Microperimetry; Diagnostic Test: M-charts

INTERVENTIONS:
Diagnostic Test: Microperimetry — Microperimetry is a procedure to assess retinal sensitivity while fundus is directly examined; it enables exact correlation between macular pathology and corresponding functional abnormality.
Diagnostic Test: M-charts — The M-chart (Inami Co., Tokyo, Japan) is a diagnostic tool developed by Matsumoto to quantify the degree of metamorphopsia in patients with macular diseases.

SUMMARY:
To examine morphological and functional results after pars plana vitrectomy (PPV) with SF6 gas tamponade due to macula-on and macula-off rhegmatogenous retinal detachment (RRD) during six months of the follow-up.

DETAILED DESCRIPTION:
Background:

To examine morphological and functional results after pars plana vitrectomy (PPV) with SF6 gas tamponade due to macula-on and macula-off rhegmatogenous retinal detachment (RRD) during six months of the follow-up.

Methods:

The study included 62 eyes that underwent successful PPV with SF6 tamponade with macula-on (34 eyes) and macula-off (28 eyes) RRD preoperatively. The best-corrected visual acuity (BCVA), Amsler test, M-charts, optical coherence tomography (OCT) and microperimetry were performed at 1, 3 and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosed macula-on and macula-off rhegmatogenous retinal detachment.

Exclusion Criteria:

* history of uveitis,
* diabetic retinopathy,
* previous vitreoretinal surgery,
* glaucoma or eye trauma,
* retinal detachment combined with macular hole or proliferative vitreoretinopathy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study included 62 eyes that underwent successful vitrectomy with SF6 tamponade with macula-on (34 eyes) and macula-off (28 eyes) RRD preoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The best-corrected visual acuity (BCVA) | 1 to 6 months
  Acuity is a measure of visual performance. The eye exam seeks to find the prescription that will provide the best corrected visual performance achievable.
Amsler test | 1 to 6 months
  The standard Amsler test performs with black lines on the white background. The Amsler grid has been used so far for the qualitative assessment of the metamorphopsia since 1947.
M-charts | 1 to 6 months
  The M-charts consist of 19 dashed lines with increasing distance between points in the range of 0.2 ° to 2.0 ° viewing angle. Matsumoto developed M-charts for quantitative metamorphopsia evaluation in macula diseases in 1990. M-charts provide more information than Amsler chart in regard to the horizontal and vertical lines.
Central retinal thickness | 1 to 6 months
  Quantitative thickness measurements derived from the "fast macular scan" algorithm report retinal thickness at several locations including the center point, central subfield, and 4 inner and 4 outer zones of the macula.
Microperimetry | 1 to 6 months
  Microperimetry is a procedure to assess retinal sensitivity while fundus is directly examined; it enables exact correlation between macular pathology and corresponding functional abnormality.

CONTACTS AND LOCATIONS:
Locations (1):
- General Department of Ophthalmology in Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: Yes
All data will be available in brief.

REFERENCES:
- [Derived] Borowicz D, Nowomiejska K, Nowakowska D, Brzozowska A, Toro MD, Avitabile T, Junemann AG, Rejdak R. Functional and morphological results of treatment of macula-on and macula-off rhegmatogenous retinal detachment with pars plana vitrectomy and sulfur hexafluoride gas tamponade. BMC Ophthalmol. 2019 May 24;19(1):118. doi: 10.1186/s12886-019-1120-3. PMID 31126280